CLINICAL TRIAL: NCT05243862
Title: Phase II Study of PolyPEPI1018 Vaccine in Combination with Atezolizumab in Participants with Relapsed or Refractory Microsatellite-stable Metastatic Colorectal Cancer.
Brief Title: Safety and Activity of PolyPEPI1018 Plus Atezolizumab in Colorectal Cancer.
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Treos Bio Limited (Industry)
Collaborators: Mayo Clinic (Other); Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OBERTO-301
Record Dates: First submitted 2022-01-26; First posted 2022-02-17 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2024-11

CONDITIONS: Colorectal Cancer Metastatic
Keywords: MSS; Peptide Vaccine; Cancer vaccine; PolyPEPI1018; Checkpoint inhibitor; PD-L1 inhibitor; Atezolizumab
MeSH Terms: interventions — atezolizumab

STUDY DESIGN:
Intervention Model Description: Following the Simon's 2-stage design, 18 participants will be enrolled in the first stage. If no participant with a response is observed, the study will be terminated for futility. If ≥ 1 participants achieve a response, then the study can proceed to the second stage, and additional 10 participants will be enrolled to the second stage.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- PolyPEPI1018 plus Atezolizumab (Experimental): Participants receive every 3 weeks PolyPEPI1018 CRC Vaccine (Emulsified solution, 0.2 mg/peptide, 6 peptides total, and Montanide™ ISA51VG adjuvant), by SC injection in combination with Atezolizumab (Injectable solution,1200mg/20mL) by IV injection.
  Interventions: Drug: PolyPEPI1018; Drug: Atezolizumab

INTERVENTIONS:
Drug: PolyPEPI1018 — PolyPEPI1018 vaccine contains 6 synthetic peptides emulsified with the adjuvant Montanide™. The peptides were selected to induce T cell responses against 12 dominant epitopes from 7 tumor-specific antigens, which are the most frequently expressed antigens in colorectal cancer.
  Other Names: PolyPEPI1018 CRC vaccine
Drug: Atezolizumab — Atezolizumab is a fully humanized, engineered monoclonal antibody of IgG1 isotype against the protein programmed cell death-ligand 1.
  Other Names: Tecentriq

SUMMARY:
This is a multicenter, open label, phase II trial to determine the safety, tolerability, and immunogenicity and initial clinical activity of the combination treatment of PolyPEPI1018 vaccine and atezolizumab in participants with MSS CRC who have progressed on 2 or 3 prior regimens.

DETAILED DESCRIPTION:
This is a multicenter, open label, phase II trial to determine the safety, tolerability, and immunogenicity and initial clinical activity of the combination treatment of PolyPEPI1018 vaccine and atezolizumab in participants with MSS CRC who have progressed on 2 or 3 prior regimens. Both agents will be administered on an every-3-week schedule until documented progression. A Simon's 2-stage design will be used for the initial assessment of efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent for the trial.
2. Adults 18 years or older on the day of signing informed consent.
3. Histologically or cytologically confirmed CRC that is metastatic.
4. Primary and/or metastatic tumor(s) that is known to be MSS as determined locally
5. Must have had 2-3 prior lines of therapy for CRC in the advanced or metastatic setting, including all of the following in the absence of contraindications: a) fluoropyrimidine, b) oxaliplatin, c) irinotecan, d) one or more biologics depending on the clinical scenario. Prior regorafenib and/or TAS-102 are allowed but not required. Note: a line of therapy is generally considered >2 weeks of exposure to the same regimen followed by radiographically documented progression. Agents that are mechanistically similar (e.g. 5-fluorouracil and capecitabine) and are used interchangeably due to tolerability but not progression may be considered as components of the same regimen upon discussion with the medical monitor.
6. Willingness to undergo biopsy prior to study therapy and after approximately 6 weeks of study therapy. If biopsy on study is not feasible, then archival tissue must be available from within 90 days of signing consent.
7. Willingness to undergo buccal swab prior to study therapy for the determination of HLA profile.
8. Documented radiographic progression after the last regimen prior to entry on this study.
9. Measurable disease, as defined by RECIST v1.1. Previously irradiated lesions can only be considered as measurable disease if disease progression has been unequivocally documented at that site since radiation.
10. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
11. Adequate organ functions as defined by the following laboratory parameters at baseline (laboratory parameters outside of these ranges that are deemed clinically insignificant should be discussed with the medical monitor):

    1. Absolute neutrophil count ≥1.5 x 109/L;
    2. Hemoglobin ≥9 g/dL: transfusion to achieve this cutoff is not allowed within 14 days of first dose of study therapy;
    3. Platelet count ≥100,000/mm3;
    4. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 x upper limit of normal (ULN) - ASL and/or ALT may be ≤5 x ULN in the setting of liver metastases;
    5. Total bilirubin ≤ 1.5 x institutional ULN;
    6. Serum creatinine within normal limits or calculated creatinine clearance >60 mL/min/1.73 m2 using the Cockroft-Gault method (Appendix 2) for participants with serum creatinine levels above or below the institutional normal range;
    7. Albumin ≥3.0 g/dL;
    8. Acceptable coagulation parameters including international normalized ratio (INR) <1.5 and partial thromboplastin time (PTT) ≤ institutional ULN in the absence of anticoagulation (participant on anticoagulants must be discussed with the medical monitor).
12. Has no major existing comorbidities or medical conditions that will preclude therapy in the view of the investigator.
13. Resolution to Grade ≤1 by the National Cancer Institute Common Terminology Criteria for Adverse Events, Version 5.0 (NCI-CTCAE v 5.0) of all clinically significant toxic effects of prior therapies (with exception of peripheral neuropathy).
14. Female participants are eligible to participate if at the time of screening are not pregnant, not breastfeeding, and at least one of the following conditions applies: (a) Not a woman of childbearing potential (WOCBP); or (b) WOCBP who (i) agrees to use highly effective contraception starting with the screening visit through 90 days after the last dose of study treatment; and (ii) must have a negative urine or serum pregnancy test within 72 hours prior to receiving any dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.

    * Childbearing potential is defined by at least one of the following: (a) ≥50 years of age and has not had menses for greater than 1 year; (b) amenorrheic for ≥2 years without a hysterectomy and bilateral oophorectomy and a follicle-stimulating hormone value in the postmenopausal range upon pre-study (screening) evaluation; (c) has had hysterectomy, bilateral oophorectomy or tubal ligation.
    * Highly effective contraception is defined in Appendix 3 or per national or local guidelines.
    * Abstinence is acceptable if this is the established and preferred method of contraception/lifestyle of the participant.
15. Male participants with a female partner(s) of childbearing potential must agree to use highly effective contraception throughout the study starting with the screening visit through 90 days after the last dose of study treatment is received by the male participant. Male participants with pregnant partners must agree to use a condom; no additional method of contraception is required for the pregnant partner.

    * Abstinence is acceptable if this is the established and preferred method of contraception of the participant.

Exclusion Criteria:

1. Prior treatment with an anti-CTLA-4, anti-PD-1, anti-PD-L1, anti-PD-L2 or any other checkpoint inhibitors.
2. Has received prior anticancer therapy (chemotherapy, targeted therapies, radiotherapy, or immunotherapy) within 28 days of the first dose of study therapy or 5 half-lives (whichever is shorter) if at least 10 days have elapsed between the last dose of such agents and the first dose of study therapy. NOTE: Patients who have been given palliative radiotherapy to peripheral sites (e.g., bone metastases) may enroll before 28 days have elapsed if they have recovered from any acute toxicities.
3. Has received a live vaccine within 28 days of the first dose of study therapy.
4. Has had major surgical procedure, open biopsy or significant traumatic injury within 28 days of the first dose of study therapy.
5. Participating in another research study involving receipt of an investigational product 21 days prior to study therapy.
6. History of autoimmune disease, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis. Note: Patients with a history of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone are eligible for this study. Patients with controlled Type I diabetes mellitus on a stable dose of insulin regimen are also eligible for this study.
7. Receiving systemic corticosteroids within one week prior to the first dose of study therapy. Exceptions: corticosteroid use as a premedication for intravenous (IV) contrast, intermittent corticosteroid use (e.g., daily prednisone at doses of ≤10 mg or equivalent), bronchodilators, inhaled steroids, or local steroid injections (except at the proposed injection site of PolyPEPI1018) are acceptable.
8. History of anaphylaxis in relation to vaccination or the administration of a protein product.
9. Has known allergy to any component of the study treatment formulation(s).
10. Has symptomatic interstitial lung disease (ILD) or ILD which may interfere with detection and management of new immune-related pulmonary toxicity.
11. Prior allogeneic bone marrow transplantation or solid organ transplant.
12. Has known, active central nervous system (CNS) metastases and/or leptomeningeal metastases. Patients with previously treated, stable CNS metastases may participate if (a) there is no evidence of progression by imaging [magnetic resonance imaging (MRI) or computed tomography (CT) as used during the prior imaging] at least 28 days prior to the first dose of study therapy; (b) resolution or return to baseline of neurologic symptoms; and (c) no requirement for steroids to manage symptoms of brain metastases for at least 28 days prior to first dose of study therapy.
13. Active infection requiring systemic therapy.
14. Significant liver cirrhosis defined as Child-Pugh Class B or C (Appendix 4).
15. Active infection with human immunodeficiency virus (HIV) except participants who are currently stable on antiretroviral therapy (ART) for at least 4 weeks and agree to adhere to ART during study therapy, have HIV viral load of <400 copies per milliliter (/mL) at screening (or undetectable per local criteria), and have CD4 T cell counts ≥200/microliter.
16. Active hepatitis B (HBV) or C (HCV) infection. For participants with evidence of HBV infection, the HBV viral load must be undetectable on suppressive therapy, if indicated. For participants with HCV, infection must have been treated and cured or participants are currently on treatment and have an undetectable HCV viral load.
17. History or evidence of cardiovascular disease, chronic respiratory disease, gastrointestinal disease, liver disease, renal disease, endocrine disorder or any other medical or psychiatric condition that in the opinion of the investigator will significantly increase the safety risk for the subject or confound the interpretation of the study data.
18. Pregnant or breast-feeding or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 90 days after the last dose of study treatment.
19. History of another active malignancy that has required therapy within 2 years prior to first dose of study therapy, except basal cell carcinoma of the skin, squamous cell carcinoma of the skin, prostate cancer or in situ cervical cancer that has undergone potentially curative therapy or is felt by the investigator to be at low risk for recurrence is allowed.
20. Substance abuse, medical, psychological or social conditions that may interfere with the subject's participation in the study or evaluation of the study results.
21. In the opinion of the investigator, participant has rapidly progressing disease, OR has life expectancy <3 months, OR would be unable to receive at least one study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2022-06-02 (Actual); Primary Completion 2024-07-08 (Actual); Study Completion 2026-06-02 (Estimated)

PRIMARY OUTCOMES:
The incidence and severity treatment related Adverse Events | From 1st dose until 90-Days after last dose
  The incidence and severity [according to the National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0 (v5.0)] of all adverse events (AEs), related AEs, all SAEs, and related SAEs
Administration safety | During the vaccine administration or within 60 minutes following administration
  Number and proportion of participants with any clinically significant change in vital signs (i.e., blood pressure, pulse rate, respiratory rate, body temperature) during the vaccine administration or within 60 minutes following administration

SECONDARY OUTCOMES:
Objective Response Rate assessment | From study entry up to 2 years
  By computed tomography (CT) scan or other appropriate radiographic imaging at Screening Visit and at specified intervals on study therapy by the investigator and per RECIST 1.1
Duration of Response assessment | From study entry up to 3 years
  DoR from the first demonstration of response per RECIST 1.1 to the first demonstration of radiographic progression per RECIST 1.1
Progression Free Survival assessment | From study entry up to 3 years
  PFS time from the first dose of study therapy to radiographic progression or death from any cause
Overall Survival assesment | From study entry up to 3 years
  OS time from the first dose of study therapy to death from any cause
PEPI Listing | 1 year
  List number of PEPIs identified by PEPI Test
Measured Effector T Cell Immune Response | From study entry up to 2 years
  Effector T cell response against vaccine antigens as measured by ex vivo interferon (IFN)-gamma Enzyme-Linked ImmunoSpot (ex vivo ELISPOT) assay at baseline and at specified intervals on study therapy
Measured Memory T Cell Immune Response | From study entry up to 2 years
  Memory T cell response against vaccine antigens of PolyPEPI1018 as measured by in vitro stimulated interferon (IFN)-gamma Enzyme-Linked ImmunoSpot (IVS ELISPOT) assay at baseline and at specified intervals on study therapy

CONTACTS AND LOCATIONS:
Overall Officials: Joleen Hubbard, MD, Principal Investigator — Mayo Clinic; Hagop Youssoufian, MD, Study Director — Treos Bio Ltd.
Locations (3):
- United States (3):
  - Mayo Clinic, Phoenix, Arizona
  - Mayo Clinic, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Evaluation of safety, immunogenicity and preliminary efficacy of PolyPEPI1018 vaccine in subjects with metastatic colorectal cancer (mCRC) with a predictive biomarker — http://doi.org/10.1093/annonc/mdz246.083
- See also: P329 PolyPEPI1018 off-the shelf vaccine as add-on to maintenance therapy achieved durable treatment responses in patients with microsatellite-stable metastatic colorectal cancer patients (MSS mCRC) — https://jitc.bmj.com/content/7/Suppl_1/282